CLINICAL TRIAL: NCT02865330
Title: Spanish Urological Association Registry of Patients on Active Surveillance
Status: Recruiting | Type: Observational
Sponsor: Fundación Instituto Valenciano de Oncología (Other)
Responsible Party: Sponsor
Other Study IDs: AEU-PIEM/2014/0001
Record Dates: First submitted 2016-06-06; First posted 2016-08-12 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: Intermediate Risk Prostate Cancer; Low Risk Prostate Cancer; Active Surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: None Retained — 7.5 ml of blood sample Biopsy sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry — National Registry of patients with prostate cancer as monitored through active surveillance, with the intention of testing the hypothesis that cancer-specific mortality in very low-risk and low-risk patients is less than 5% at 15 years.

SUMMARY:
Description:

Multicentre observational study, not randomized. Ambispective character (retro and prospective). Opened to any member of the Asociación Española de Urología (AEU), public and private medicine.

Justification:

Active surveillance is a strategy proposed to control the overtreatment derived from the opportunist screening in prostate cancer (PCa).

Its development in our country is erratic and different in every Center. This database tries to include most of patients included in active surveillance in Spain with a few minimal inclusion criteria.

Multicentre registry and follow up of the active surveillance in Spain.

Hypothesis:

Mortality cancer specific for PCa includible in active surveillance to 15 years is lower than 5 %.

ELIGIBILITY:
Inclusion Criteria:

1. PSA ≤ 10 ng / mL; if prostate volume> 60 cc in transrectal, ultrasound includable with PSA>10 ng / ml if PSAD <0.20
2. Local Stadium DRE; cT1c -cT2a
3. Diagnosis of transrectal ultrasound guided biopsy minimum 10 cylinders
4. Adenocarcinoma Prostate Gleason ≤ 6 (3 + 3) with local and central pathology review
5. Maximum number of cylinders = 2 and none of them more than 5mm tumor or more than 50% of assignment
6. <80 years and greater expectancy to 10 years life (Charlson score)
7. Patients able to understand active surveillance and sign the Informed Consent

Exclusion Criteria:

1. Patient not be able to accept up with repeat biopsies
2. Patient who does not want to sign the Informed Consent
3. Hospital where the possibility of a biopsy confirmation at 6 months is not guaranteed under the terms of the inclusion criteria
4. Patients with a history of ASAP (atypical small acinar proliferation or atypical microglands)
5. Patients with treatment with inhibitors of 5-alpha-reductase as dutasteride (Avidart®) and finasteride (Proscar®) during the previous six months
6. Patients who have undergone during the 6 months prior to any treatment symptomatic benign prostate hyperplasia, or any invasive urological procedure. It can be associated with an increase of PSA prior to phlebotomy. These therapies include, but they are not limited to, prostate biopsy, thermotherapy, microwave therapy, laser, urethral resection of the prostate, urethral catheterization and the lower genitourinary tract endoscopy.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spain male residents diagnosed with low risk PCa (NCCN)
Sampling Method: Non-Probability Sample
Enrollment: 946 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-06 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
Cancer specific survival in patients in active surveillance | up to 15 years
  Global CSS will be recorded, independently of each Center protocol, from enrollment to death due to PRostate Cancer Estimated CSS will be analyzed at 5, 10 and 15 years from initiation of the protocol.
  To this purpose, patients will be followed although they progressed and went into active treatment.
Overall survival | Date randomization-date death, or up to 15 years, whichever came first
  Global OS will be recorded, independently of each Center protocol, from enrollment to death of any cause Estimated OS will be analyzed at 5, 10 and 15 years from initiation of the protocol To this purpose, patients will be followed although they progressed and went into active treatment or if the kept in active surveillance till their death due to any cause.
Active treatment-free interval | Date start active surveillance-stop active surveillance due to active treatment, or up to 15 years, whichever came first
  Time to active treatment will be recorded, independently of each Center protocol, from enrollment to any other active due to prostate cancer progression or patient desire to receive any active treatment Estimated active treatment free survival will be analyzed at 2, 5 and 10 years from initiation of the protocol.
Characterization of pathologically agressive tumors by Gleason score | From the study start and stop until 15 years
  Characterization of pathologically agressive tumours will be done by analyzing the pathological reports of radical prostatectomy specimens derived from patients included in the protocol that went on to radical prostatectomy. This has no time frame, although time of radical prostatectomy will be a variable to take in account for comparisions among different timings of performace of radical prostatectomies.
Characterization of pathologically agressive tumors by TNM | From the study start and stop until 15 years
  Characterization of pathologically agressive tumours will be done by analyzing the pathological reports of radical prostatectomy specimens derived from patients included in the protocol that went on to radical prostatectomy. This has no time frame, although time of radical prostatectomy will be a variable to take in account for comparisions among different timings of performace of radical prostatectomies.

SECONDARY OUTCOMES:
Quality of Life in patients with active surveillance | up to 5 years
  Assessed with CAVIPRESS-30 questionaires
Quality of Life in patients with active surveillance | up to 5 years
  Assessed with EPIC-20 questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Jose Rubio Briones, MD, PhD, Principal Investigator — IVO; Ángel Borque Fernando, MD, PhD, Principal Investigator — Hospital Miguel Servet
Locations (1):
- Instituto Valenciano de Oncología, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rubio-Briones J, Borque A, Esteban LM, Iborra I, Lopez PA, Gil JM, Pallas Y, Fumado L, Martinez-Breijo S, Chantada V, Gomez E, Quicios C, Congregado CB, Medina R, Ortiz M, Montesino M, Clar F, Soto J, Campa JM. Preliminary results of the Spanish Association of Urology National Registry in Active Surveillance for prostate cancer. Actas Urol Esp. 2016 Jan-Feb;40(1):3-10. doi: 10.1016/j.acuro.2015.05.006. Epub 2015 Jun 23. English, Spanish. PMID 26115777
- [Background] Borque-Fernando A, Rubio-Briones J, Esteban LM, Collado-Serra A, Pallas-Costa Y, Lopez-Gonzalez PA, Huguet-Perez J, Sanz-Velez JI, Gil-Fabra JM, Gomez-Gomez E, Quicios-Dorado C, Fumado L, Martinez-Breijo S, Soto-Villalba J. The management of active surveillance in prostate cancer: validation of the Canary Prostate Active Surveillance Study risk calculator with the Spanish Urological Association Registry. Oncotarget. 2017 Oct 24;8(65):108451-108462. doi: 10.18632/oncotarget.21984. eCollection 2017 Dec 12. PMID 29312542
- [Derived] Rubio-Briones J, Borque-Fernando A, Esteban Escano LM, Wong A, Guijarro Cascales A, Gomez Gomez E, Gil Fabra JM, Sanguedolce F, Gomez-Veiga F, Lopez Gonzalez PA, Plata Bello A, Rodriguez Garcia N, Montesino Semper M, Suarez Novo JF, Hajianfar R, Fumado Ciutat LL, Gonzalez Alfaro A, Duarte Ojeda JM, Bono Arino A, Quicios Dorado C, Loizaga Iriarte A, Garcia Fadrique G, Gimenez Bachs JM, Garcia Barreras S, Pallas Costa Y, Vilaseca Cabo A, Rodrigo Aliaga M, Campanario Perez F, Servian P, Campa Bortolo JM, Soto Delgado M, Rodriguez de Ledesma JM, Sanchez Rodriguez C, Chantada Abal V, Hernandez Martinez YE, Herrera Imbroda B, Dolezal P, Gual Frau J, Medrano Llorente P, Moreno Jimenez J, Serrano Uribe JS, Congregado Ruiz CB, Reyes A, Fernandez Aparicio T, Garcia Rodriguez J, Cuadras Sole M, Garcia Segui A, Pacheco Bru JJ, Mayor de Castro J, Mira Moreno A, Molina Suarez JL. Real World Evidence of Active Surveillance for Prostate Cancer in Spain; Midterm Results. Cancer Med. 2025 Sep;14(17):e71173. doi: 10.1002/cam4.71173. PMID 40926355
- [Derived] Borque-Fernando A, Rubio-Briones J, Esteban LM, Dong Y, Calatrava A, Gomez-Ferrer A, Gomez-Gomez E, Gil Fabra JM, Rodriguez-Garcia N, Lopez Gonzalez PA, Garcia-Rodriguez J, Rodrigo-Aliaga M, Herrera-Imbroda B, Soto-Villalba J, Martinez-Breijo S, Hernandez-Canas V, Soto-Poveda AM, Sanchez-Rodriguez C, Carrillo-George C, Hernandez-Martinez YE, Okrongly D. Role of the 4Kscore test as a predictor of reclassification in prostate cancer active surveillance. Prostate Cancer Prostatic Dis. 2019 Mar;22(1):84-90. doi: 10.1038/s41391-018-0074-5. Epub 2018 Aug 14. PMID 30108375
- See also: Enlace a la página web de la asociación Española de Urología — http://piem.aeu.es/proyectos/VACP/